CLINICAL TRIAL: NCT01345981
Title: A Comparison of Pain Severity on Injection of MCT/LCT Propofol Between Lidocaine 20 mg, 40 mg, and Without Lidocaine.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Assistant Professor Nalinee Kovitwanawong, Department of Anesthesiology Faculty of Medicine Prince of Songkla University Thailand
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: propofol-pain
Record Dates: First submitted 2011-04-25; First posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Adult Disease
MeSH Terms: conditions — Disease | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- lidocaine 20 mg (Experimental): intravenous lidocaine
  Interventions: Drug: Lidocaine
- lidocaine 40 mg (Experimental): intravenous lidocaine 40 mg
  Interventions: Drug: Lidocaine
- normal saline (Placebo Comparator): 2 ml
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — dosage 20 mg and 40 mg

SUMMARY:
To compare the severity of pain on injection of MCT/LCT propofol with lidocaine 20 mg, 40 mg, and without lidocaine.

DETAILED DESCRIPTION:
Background: Intravenous injection of propofol produces pain. Many factors are involved and various techniques have been tried to minimize the propofol-induce pain with variable results.

Objective: To compare the severity of pain on injection of MCT/LCT propofol with lidocaine 20 mg, 40 mg, and without lidocaine.

Design: Randomize controlled trial. Method: Two hundred and ten ASA class I - III patients undergoing elective surgery were blinded and equally allocated into 3 groups. Patients in group N, L1, and L2 received MCT/LCT propofol 10 ml mixed with 0.9% NaCl 2 ml, 1% lidocaine 2 ml, and 2% lidocaine 2 ml respectively. Pain at time of propofol injection was assessed by blinded anesthesiologist on a four point scale ; 0 = no pain, 1 = mild pain, 2 = moderate pain, and 3 = severe pain. Results: Patient's demographic data of each group were similar. There were significant differences in the incidence of propofol injection without pain among groups (p<0.001). The numbers of patients who had moderate and severe pain in groups L1 and L2 were significantly less than those in group N (p<0.001). The mean blood pressure and heart rate were not significant differences in among groups. Conclusion : The amount of 20 mg, and 40 mg lidocaine to MCT/LCT propofol in our study is equally effective in decreasing pain and more effective than MCT/LCT propofol alone group significantly. They were no significant differences in hemodynamics change in among groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I - III patients
* undergoing elective surgery
* age 18-75 years

Exclusion Criteria:

* allergy to propofol and lidocaine
* abnormal liver and renal functions
* has psychological problem or drug abuse
* has recieved analgesic drug 2 weeks prior to surgery
* risk of aspiration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
pain on injection | 30 minutes
  4 points score for pain:o=no pain,1=mild pain,2=moderate pain,3=severe pain after propofol injection

SECONDARY OUTCOMES:
hemodynamic change | 30 minutes
  blood pressure and heart rate after propofol injection

CONTACTS AND LOCATIONS:
Locations (1):
- Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand